CLINICAL TRIAL: NCT02351141
Title: Structure and Function MRI of Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Grace Parraga (Other)
Responsible Party: Sponsor-Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ROB0037
Record Dates: First submitted 2015-01-15; First posted 2015-01-30 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Asthma
Keywords: Noble Gas MRI; Pulmonary Function; Quality of Life Questionnaires
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asthma Patients (Other): All enrolled asthma patients will undergo hyperpolarized noble gas MRI with Helium-3 and/or Xenon-129, Pulmonary Function Tests, Quality of Life Questionnaires, dyspnea scales in two visits over three years.
  Interventions: Other: Hyperpolarized Noble Gas MRI

INTERVENTIONS:
Other: Hyperpolarized Noble Gas MRI — Hyperpolarized Helium-3 and/or Xenon-129. Noble gas magnetic resonance imaging (MRI) has recently emerged as another research approach for the non-invasive measurement of lung structure and function, including conduction of gas through airways and into airspaces.
  Noble gas MRI provides a complimentary and alternative method for evaluating lung disease and may be superior to CT because it allows simultaneous visualization of both airway and airspace structure and function.

SUMMARY:
The investigators will apply 129Xenon and/or 3He image acquisition and analysis methods in 200 asthma patient volunteers in order to characterize and probe the relationship between lung structure and function using imaging.

DETAILED DESCRIPTION:
This is an exploratory, longitudinal study with no medication evaluated. 200 asthma patients will visit the Clinical Imaging Research Laboratories at Robarts Research Institute two times over three years: at baseline, and at three years. For the first 60 subjects there will be 3 additional visits - two visits within 4 weeks of baseline (BL+2 weeks; BL+4 weeks; BL+78 weeks) in order to help generate reproducibility data and temporal maps.

For all subjects, the Baseline visit will include 129Xe and/or 3He MRI, chest CT, sputum induction, Pulmonary Function Tests, Airwave Oscillation test, Lung Clearance Index test, BORG Dyspnea Scale, and MRC Dyspnea Scale. All procedures will be before, during and after methacholine challenge (MCh). For V2, all but CT and MCh will be acquired.

Visits 1a and 1b will include MRI, Pulmonary Function Tests including Airwave Oscillation and Lung Clearance Index, and dyspnea questionnaires; Visit 1c will also include sputum induction.

There will be a telephone call at 52+/- 2 weeks, and 104 +/- 2 weeks. to track exacerbations and update medications. Subjects will complete self-assessments in the form of a) the Asthma Quality of Life Questionnaire with Standardized Activities (AQLQ(S)) bi-weekly, and the Asthma Control Diary (weekly) between visits. Self-reported data (the weekly asthma control diary and bi-weekly AQLQ(S)) will be uploaded by each subject monthly to the investigators website using a confidential and password protected upload (www.imaging.robarts.ca/~gep/ForPatients.htm).

ELIGIBILITY:
Inclusion Criteria:

* Subjects male and female aged 18-60 with a clinical diagnosis of asthma
* Smoking history ≤ 1 pack/year
* Subject understands the study procedures and is willing to participate in the study as indicated by signature on the informed consent
* Subject is judged to be in otherwise stable health on the basis of medical history
* Subject able to perform reproducible pulmonary function testing (i.e., the 3 best acceptable spirograms have FEV1 values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater.)
* FEV1 >60% predicted

Exclusion Criteria:

* Patient is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material
* Patient is unable to perform spirometry or plethysmography maneuvers
* Subject has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants.) (At the discretion of the MRI Technologist/3T Manager)
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.
* Patient is pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Ventilation Defect Percent as measured by Xenon-129 and/or Helium-3 MRI | 3 years
  VDP is a widely used noble gas MRI biomarkers that is calculated by normalizing ventilation defect volume to the thoracic cavity

SECONDARY OUTCOMES:
Forced Expiratory Volume (FEV1) measured by spirometry | 3 years
  The volume of air that is exhaled in the first second is referred to as FEV1
Additional Pulmonary Function measurements | 3 years
  Measurements include Functional Residual Capacity (FRC); Total Lung Capacity (TLC); Inspiratory Capacity (IC); Airway Resistance (Raw); Forced Vital Capacity (FVC); FEV1/FVC Ratio
Quality of Life questionnaires | 3 years
  questionnaires
Dyspnea Scale | 3 years
  Scale

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] McIntosh MJ, Kooner HK, Eddy RL, Wilson A, Serajeddini H, Bhalla A, Licskai C, Mackenzie CA, Yamashita C, Parraga G. CT Mucus Score and 129Xe MRI Ventilation Defects After 2.5 Years' Anti-IL-5Ralpha in Eosinophilic Asthma. Chest. 2023 Jul;164(1):27-38. doi: 10.1016/j.chest.2023.02.009. Epub 2023 Feb 11. PMID 36781102
- [Derived] Capaldi DPI, Guo F, Xing L, Parraga G. Pulmonary Ventilation Maps Generated with Free-breathing Proton MRI and a Deep Convolutional Neural Network. Radiology. 2021 Feb;298(2):427-438. doi: 10.1148/radiol.2020202861. Epub 2020 Dec 8. PMID 33289613
- [Derived] Eddy RL, Svenningsen S, Kirby M, Knipping D, McCormack DG, Licskai C, Nair P, Parraga G. Is Computed Tomography Airway Count Related to Asthma Severity and Airway Structure and Function? Am J Respir Crit Care Med. 2020 Apr 15;201(8):923-933. doi: 10.1164/rccm.201908-1552OC. PMID 31895987